CLINICAL TRIAL: NCT04363788
Title: Should we Use Double Gloves During Procedures With Suspected/Confirmed COVID-19 Patient?
Brief Title: Needle Stick Injuries in Emergency Medical Service Practice
Status: Completed | Type: Observational
Sponsor: Lazarski University (Other)
Collaborators: Medical University of Bialystok (Other); Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: OH_PPE_1
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Cardiac Arrest; Needle Stick; Injuries; Glowe
Keywords: needle stick injuries; SARS-CoV-2; COVID-19; personal protective equipment; paramedic; emergency medical service
MeSH Terms: conditions — Heart Arrest; Needlestick Injuries; Wounds and Injuries; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiopulmonary resuscitation: The study was based on dying gloves used during resuscitation. The gloves were secured with disposable hermetically sealed pouches and described by one of the EMS team members - each time after resuscitation was completed.
  Interventions: Procedure: double gloves

INTERVENTIONS:
Procedure: double gloves — The study was based on dying gloves used during resuscitation. The gloves were secured with disposable hermetically sealed pouches and described by one of the EMS team members - each time after resuscitation was completed.
  Other Names: DL

SUMMARY:
During the pandemic era, medical personnel should wear full protective suits. However, they limit the performance of medical procedures. One of the main questions is whether to use double gloves. The study was based on dying gloves used during resuscitation. The gloves were secured with disposable hermetically sealed pouches and described by one of the EMS team members - each time after resuscitation was completed.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* Medical profession (paramedics, nurses, physicians) working in Emergency Medical Service

Exclusion Criteria:

* Not meet the above criteria
* Wrist or low back diseases

Age Groups: Child, Adult, Older Adult
Study Population: Medical profession (paramedics, nurses, physicians) working in Emergency Medical Service performing prehospital advance life support
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Number of visible puncture | 1 day
  visible puncture

SECONDARY OUTCOMES:
WLT | 1 day
  Water leak test was used to checking unnoticed gloves damage

CONTACTS AND LOCATIONS:
Locations (1):
- Lazarski Univeristy, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
data will be part of manuscript